CLINICAL TRIAL: NCT06152302
Title: Analysis of Mobility in the Bath for Infants Affected With Spinal Muscular Atrophy
Brief Title: Test of Aquatic Mobility of SMA Infants
Acronym: BAINSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP231293; 2022-A01419-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-10-30; First posted 2023-11-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Infantile Spinal Muscular Atrophy
Keywords: SMA; infantile; bath test; water mobility test; inertial sensors; floppy infant; Garches
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscle Hypotonia

STUDY DESIGN:
Intervention Model Description: There is one arm in this study, without comparator group.
  The comparison will be between data of movements in the outside water condition and data of inside water condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobility Assessment (Experimental): This study involves a single arm, without a comparator group. The comparison will be made between the data for movements in conditions outside the water and inside the water.
  Interventions: Other: Mobility study in dry conditions; Other: Mobility study in water conditions

INTERVENTIONS:
Other: Mobility study in dry conditions — Record the movements of the baby's extremities using inertial sensors while the baby moves outside of the water.
Other: Mobility study in water conditions — Record the movements of the baby's extremities using inertial sensors while the baby moves inside the water.
  Other Names: Garches Bath Test (GBT)

SUMMARY:
Spinal muscular atrophy (SMA) is a genetic neurodegenerative disease impacting spinal cord motor neurons, leading to motor and respiratory issues and, ultimately, death. With emerging therapies, a need arises to enhance motor function assessment in severely hypotonic infants (SMA type 1) as traditional scales on examination tables lack completeness due to gravity's influence.

The study team has developed a "bath test" to observe infants' motor skills in water, eliminating gravity's effects. This test aims to detect subtle movements using inertial sensors, potentially revealing more active motor neurons in aquatic conditions. It aids in identifying infants with motor improvement potential, even if they show limited mobility outside water, and tracks disease progression and therapy responses.

Presently, pediatric neurologists in France use parent-provided bathing videos for evaluations, but these lack standardization and precision. The study aims to establish a standardized evaluation protocol with quantifiable data.

The study's key objective is to evaluate severely hypotonic SMA infants using inertial sensors, including accelerometers, gyrometers, and magnetometers. The study will conduct "dry" and "water" assessments using a specially designed bathtub. This method's goal is to quantify water-based movements accurately.

Simultaneously, the study seeks to establish semi-quantitative evaluation criteria to create a clinical assessment scale for infant motor function in bathtubs. This scale will aid doctors in therapeutic decisions. The study will not influence the treatment or therapeutic decisions made for the children being tested.

Collected data from "dry" and "water" conditions will be statistically analyzed and compared to reference motor assessment scales (e.g., CHOP INTEND and HINE) and electromyography (CMAP-EMG) results, commonly used in diagnosis and monitoring. Blurred video recordings will assist in protocol monitoring and sensor data analysis.

DETAILED DESCRIPTION:
This is a multicenter research project coordinated by the Child Neuromuscular Unit at Raymond Poincaré Hospital. Additionally, two other pediatric neurology departments, part of the national neuromuscular network FILNEMUS (https://www.filnemus.fr/), will participate in the study: Necker Children's Hospital and Armand Trousseau Hospital.

The study's population will include all infants diagnosed with spinal muscular atrophy (SMA), specifically SMA type 1, who have onset before 6 months of age and have been evaluated by the French Therapeutic Commission. Participation in the study will be contingent on parental or guardian consent during follow-up visits.

Spinal muscular atrophy is a genetic neurodegenerative condition that affects spinal motor neurons, causing motor and respiratory paralysis and ultimately leading to death. As groundbreaking therapies emerge, there's an increasing need to refine the methods used to assess motor function, especially in infants with severe hypotonia due to SMA type 1. Traditional reference scales used on examination tables are limited in their accuracy because of gravitational effects. Consequently, there's growing interest in evaluating these children's motor skills in water to detect movements unburdened by gravity. Pediatric neurologists in France (SFNP) have already acknowledged the potential value of parental video recordings during infant baths. However, the lack of standardization in recording conditions, coupled with the subjective nature of video interpretations, underscores the necessity for a more standardized and quantifiable approach. Herein lies the application of our proposed evaluation utilizing inertial sensors.

Utilizing inertial sensors to detect subtle movements can highlight still-active yet minimally functional motor neurons. Such detection can be pivotal in identifying children who, despite severe motor skill limitations in traditional settings, still possess developmental potential. Our study seeks to leverage these sensors-equipped with accelerometers, gyroscopes, and magnetometers-to carry out evaluations both in ''dry'' conditions and ''water'' conditions, using a specially designed, secure bathtub.

The study aims to validate the relevance of quantifying movements in aquatic settings using inertial sensors, in order to assess motor function in very hypotonic children. Additionally, this study will contribute to the development of a semi-quantitative clinical evaluation grid for assessing infant motor function in water, assisting physicians in making more informed therapeutic decisions for these children. Data obtained from measurements with inertial sensors in both environments ("dry" and "water") will be correlated with scores from validated motor scales (CHOP INTEND; HINE-2) and the clinical characteristics of the patients (e.g., age, disease duration, SMA type, SMN2 copies, severity, CMAPs [EMG]). Anamnestic, clinical and inertial data will be anonymized.

The equipment required for the protocol comprises an examination table, a bath, a support for the head and back (https://www.neut.fr/fr/), 8 CE-validated Xsens DOT© inertial sensors, a dedicated research smartphone with the Xsens DOT© application for data export, a camera mounted on a pole connected to an acquisition tablet. The study will utilize a fixed PC computer with secure access, located in a dedicated research room within the Pediatric Neurology and Intensive Care Unit at Raymond Poincaré Hospital.

Video recording throughout the evaluation will be carried out from an overhead perspective, capturing all four limbs in the frame and ensuring that the child occupies approximately 50% of the camera's field of vision. To comply with privacy regulations (MR-001), the videos will obscure any identifying features, such as faces or other body parts of the patients. These videos will serve as a reference for controlling and validating the data collected by the inertial sensors.

The study's outputs will include inertial data from 8 inertial sensors placed on the arms (2), forearms (2), thighs (2), and legs (2). Our motor evaluation process is split into two distinct phases, totaling 6 minutes: a "dry" phase affected by gravity, and a "water" phase where gravity's effects are mitigated. The surrounding time is allocated for essential tasks such as positioning the child, fitting the sensors, and ensuring the infant's comfort throughout the process. Notably, our study doesn't seek to alter the standard care or therapeutic decisions for the participants.

The measurements will follow a specific process:

* "Dry" phase: This involves evaluating limb movements under the constraints of gravity. The child is placed in a supine position on the examination table set horizontally (0°). To minimize signal artifacts, physical contact with the child should be avoided. If the child's behavior is unfavorable (e.g., crying), the measurement is paused and resumed once the child's condition stabilizes. Spontaneous or induced movements are collected for 2 minutes, with the entire duration filmed for monitoring the inertial sensor data.
* Intermediate phase: The diaper is removed, and the child is positioned in a support inclined at 20°, then transferred to the bathtub. This transition should be made in a reassuring manner for the child, respecting their pace of adaptation.
* "Water" phase: This phase involves evaluating limb movements without gravity constraints. Spontaneous or induced movements are collected for 4 minutes, with the entire duration filmed for monitoring the inertial sensor data. Measurements may also be paused and resumed based on the child's behavior.

The processes of sensor installation and sensor removal are accompanied by sensorimotor stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Infants with muscle weakness (commonly referred to as floppy babies):

  * Confirmed diagnosis of SMA through gene mutation or deletion (SMN1 gene).
  * Receiving standard care.
  * Age less than 12 years and a height of less than 90 cm at the time of inclusion.
* Patients enrolled in a social security scheme.
* Informed consent signed by both parents of the child and the investigator.

Exclusion Criteria:

* Patients presenting with lesions in the spinal cord or conditions affecting the cardiorespiratory system.
* Patients covered under the French Aid in Health for Foreign People program (AME).

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Delta of 95th percentile of free acceleration norm (in m/s²) | through study completion, an average of 15 months
  Difference of free acceleration norm (in m/s²) for each measurement point respectively (elbows; wrists; knees; ankles), between "dry" and "water" condition.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Quijano-Roy, MD, PhD, Principal Investigator — Paediatric neurological and intentive care unity, Raymond Poincaré Hospital - APHP; Nour Maalouf, Psychomotor Therapist DE, Study Director — Paediatric neurological and intentive care unity, Raymond Poincaré Hospital - APHP
Locations (1):
- Infantile neuromuscular unity - Department of paediatric neurological care and intentive care unity, Raymond Poincaré Hospital - APHP, Garches, France